CLINICAL TRIAL: NCT04458285
Title: A Multi-center, Randomized, Open-label, Active-controlled, 12-week Study to Evaluate the Efficacy and Safety of Sacubitril/Valsartan in Maintenance Hemodialysis Patients With Heart Failure
Brief Title: Efficacy and Safety of Sacubitril/Valsartan in Maintenance Hemodialysis Patients With Heart Failure
Acronym: ESARHD-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, ShuangXin Liu, Chief Physician, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20191025
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-07

CONDITIONS: Hemodialysis Complication; Heart Failure
Keywords: Sacubitril/valsartan; valsartan; Hemodialysis; Heart failure
MeSH Terms: conditions — Heart Failure | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril/valsartan (Experimental): Patients in experimental group will receive sacubitril/valsartan with the recommended starting dose: 50mg twice daily (if previous angiotensin converting enzyme inhibitor(ACEI), ensure 36-hour washout period), after 2-4 weeks, the dose will be doubled to the target maintenance dose of 100mg twice daily(if tolerated) for 12 weeks.
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet [Entresto]
- Valsartan (Active Comparator): Patients in active comparator group will receive Valsartan with an dose of 80 mg once daily.
  Interventions: Drug: Valsartan 80mg Tablet

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet [Entresto] — Patients in experimental group will receive sacubitril/valsartan with the recommended starting dose: 50mg twice daily (if previous ACEI, ensure 36-hour washout period), after 2-4 weeks, the dose will be doubled to the target maintenance dose of 100mg twice daily(if tolerated) for 12 weeks.
  Other Names: LCZ696 100 mg tablet
  Arms: Sacubitril/valsartan
Drug: Valsartan 80mg Tablet — Patients in active comparator group will receive Valsartan with an dose of 80 mg once daily.
  Arms: Valsartan

SUMMARY:
Sacubitril/valsartan reduces the risk of cardiovascular mortality among patients with heart failure with reduced ejection fraction, and has been recently indicated as a new treatment option with a strong level of recommendation (class I, level of evidence B) in the main international guidelines. Cardiovascular disease (CVD) is the most common cause of death in end stage renal disease (ESRD) patients undergoing hemodialysis (HD). Hence, treatments to improve mortality and specifically cardiovascular outcomes in this population are greatly needed. So far, no data available about the efficacy and safety of sacubitril/valsartan in ESRD patients undergoing hemodialysis, although this medication was noted to be effective and comparably well tolerable in those with estimated glomerular filtration rate(eGFR) 20 to 60 mL/min/1.73 m2 in the United Kingdom Heart and Renal Protection-III trial.

The purpose of this open label, randomized controlled study with prospective data collection is to assess the efficacy and safety of sacubitril/valsartan in maintenance hemodialysis patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained before any study assessment is performed.
* End stage renal disease (ESRD) patients (eGFR<15ml/min/1.73m² as measured by the Chronic Kidney Disease Epidemiology Collaboration formula at screening) who have been receiving hemodialysis 3 times a week for at least 12 weeks before registration.
* Chronic heart failure (NYHA class ≥ II) with reduced ejection fraction, defined as known LVEF ≤ 50%.
* Mean sitting systolic blood pressure(msSBP)≥110 mmHg.
* Use of angiotensin-converting enzyme inhibitors/angiotensin receptor blocker for at least 2 weeks.
* Good compliance.

Exclusion Criteria:

* Acute renal failure with hemodialysis.
* Isolated right heart failure owing to pulmonary disease, primary cause of dyspnea due to noncardiac, non-HF causes such as acute or chronic respiratory disorders.
* Systolic blood pressure lower than 100 mmHg at screening (<95 mmHg at the randomization visit).
* Previous history of intolerance to recommended target doses of angiotensin receptor blockers.
* Significant laboratory abnormalities at screening interfering with assessment of study drug safety or efficacy (such as serum potassium>5.5 or <3.5mmol/L, serum sodium<130mmol/L or alanine aminotransferase or aspartate aminotransferase>2 times the upper limit of the normal range)
* History of hypersensitivity to any of the study drugs or their excipients or to drugs of similar chemical classes.
* History of angioedema.
* Any medications that have potential for drug-drug interaction with LCZ696 will not be allowed during the study.
* Pregnant female.
* Use of sacubitril/valsartan prior to week-2.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 12 weeks
  Change from baseline in left ventricular ejection fraction (LVEF) between baseline and end of study

SECONDARY OUTCOMES:
N terminal pro B type natriuretic peptide (NT-prpBNP) | 12 weeks
  Blood samples will be collected for analysis of concentration of N terminal pro B type natriuretic peptide (NT-proBNP) every 2 weeks.
Left ventricular end diastolic volume (LVEDV) | 12 weeks
  LVEDV is measured as baseline and after 12 weeks follow-up.
Left atrial volume (LAV) | 12 weeks
  LAV is measured as baseline and after 12 weeks follow-up.
The ratio of mitral early diastolic blood flow peak and mitral annulus velocity (E/E') | 12 weeks
  E/E' is measured as baseline and after 12 weeks follow-up.
Pulmonary Artery Pressure | 12 weeks
  Pulmonary Artery Pressure is measured as baseline and after 12 weeks follow-up.
Concentration of high-sensitivity serum troponin T | 12 weeks
  Blood samples will be collected for analysis of concentration of serum troponin every 4 weeks.
NYHA functional classification | 12 weeks
  NYHA functional classification is assessed from baseline and 12 weeks follow-up.
Minnesota Heart Failure Quality of Life Questionnaire (LiHFe) | 12 weeks
  Change in health status is assessed using the disease-specific Minnesota Heart Failure Quality of Life Questionnaire.
Systolic and diastolic blood pressure | 12 weeks
  Systolic and diastolic blood pressure will be measured every 2 weeks.
Concentration of postassium | 12 weeks
  Blood samples will be collected for analysis of concentration of postassium every 2 weeks.
Electrocardiogram(ECG) | 12 weeks
  ECG QT Interval analysis was performed at baseline and 12 weeks follow-up.
Estimated glomerular filtration rate(eGFR) | 12 weeks
  Change in estimated glomerular filtration rate(eGFR)
Incidence of Angioedema | 12 weeks
  Incidence of Angioedema during the study period 12 weeks.
Concentration of alanine aminotransferase or aspartate aminotransferase | 12 weeks
  Blood samples will be collected for analysis of concentration of alanine aminotransferase or aspartate aminotransferase every 2 weeks.

OTHER OUTCOMES:
Neprilysin | 12 weeks
  The concentration of Neprilysis is measured by Human Neprilysin ELISA Kit as baseline and after 12 weeks follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Shuangxin Liu, Doctor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Haynes R, Judge PK, Staplin N, Herrington WG, Storey BC, Bethel A, Bowman L, Brunskill N, Cockwell P, Hill M, Kalra PA, McMurray JJV, Taal M, Wheeler DC, Landray MJ, Baigent C. Effects of Sacubitril/Valsartan Versus Irbesartan in Patients With Chronic Kidney Disease. Circulation. 2018 Oct 9;138(15):1505-1514. doi: 10.1161/CIRCULATIONAHA.118.034818. PMID 30002098
- [Background] Velazquez EJ, Morrow DA, DeVore AD, Duffy CI, Ambrosy AP, McCague K, Rocha R, Braunwald E; PIONEER-HF Investigators. Angiotensin-Neprilysin Inhibition in Acute Decompensated Heart Failure. N Engl J Med. 2019 Feb 7;380(6):539-548. doi: 10.1056/NEJMoa1812851. Epub 2018 Nov 11. PMID 30415601